CLINICAL TRIAL: NCT05121662
Title: Immunogenicity of COVID-19 Vaccines in MS Patients on B-cell Depleting Therapy
Brief Title: COVID-19 Vaccine Biomarker Study in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAT7220
Record Dates: First submitted 2021-11-12; First posted 2021-11-16 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; COVID-19
Keywords: Vaccine
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Multiple Sclerosis (MS): Individuals with MS on B-cell depleting therapy, non-cell depleting therapy, or no therapy.

SUMMARY:
SARS CoV-2 is the virus responsible for the pandemic COVID-19, which has resulted in nearly five million deaths worldwide since its spread in the beginning of 2020. In the United States, there are now two emergency use authorized vaccines that make use of messenger ribonucleic acid (mRNA) based technology that are highly effective for preventing COVID. However, because multiple sclerosis is an autoimmune condition, many individuals with multiple sclerosis take medicines that affect the immune system. The investigators are not sure whether individuals on certain MS medications, including medications that lower a type of immune cell called B lymphocytes, will form as robust of a response to the vaccines. In this study, the investigators will be gathering more information about effectiveness of these vaccines and bloodwork that looks at antibodies and other markers of vaccine response and by asking patients about COVID-19 infections.

DETAILED DESCRIPTION:
SARS CoV-2 is the virus responsible for the pandemic COVID-19, which has resulted in nearly five million deaths worldwide since its spread in the beginning of 2020. In the United States, there are currently two emergency use authorized mRNA based vaccines against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Multiple sclerosis (MS) is a neurological autoimmune disease involving the central nervous system and requiring long-term immunomodulating therapy to control relapse and progression. While there are many approved medications for the treatment of MS, agents that work through B-lymphocyte depletion or sequestration are among the commonly used treatments. There is concern that individuals with low levels of circulating B-cells might not mount an effective humoral or cellular immune response after vaccination. Moreover, it remains to be understood whether, at certain timepoints within the treatment cycle, there is a greater immune response mounted while on B-cell depleting medication. Availability of such knowledge could guide counseling and management of patients on immunomodulatory therapy. Aim: To ascertain efficacy of mRNA based SARS CoV-2 vaccines in individuals with MS across the immunotherapy spectrum, via biomarker data of humoral and cellular immunity and via clinical data. Blood will be drawn for markers of immunity and sequence-based analysis before and after vaccination at predetermined time points. The investigators will document the type of immunotherapy being used at the time of vaccination. Clinical data on diagnosis of SARS-CoV2 infection will be collected at each of the prespecified timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any form of multiple sclerosis based on 2017 McDonald Criteria
* Ages 18 to 70
* No history of prior vaccination against SARS-CoV-2 at the start of the study

Exclusion Criteria:

* Unable to obtain blood draws at predetermined time points
* Pregnant at time of enrollment or planning pregnancy during upcoming 6 month period after vaccination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with multiple sclerosis who received vaccination 50 of these subjects will be on B-cell depleting agents (ofatumumab, ocrelizumab, and rituximab) and the other 50 will either not be on immunotherapy for MS or will be on non-cell depleting therapies (glatiramer acetate, beta-interferons, natalizumab, dimethyl fumarate, diroxyl fumarate, teriflunomide, siponimod, fingolimod and ozanimod).
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Level of Receptor Binding Domain (RBD) | Up to 24 months
  Level of RBD binding Immunoglobulin G (IgG) in blood samples

SECONDARY OUTCOMES:
Level of SARS-CoV-2 Neutralizing Antibodies | Up to 24 months
  Level of SARS-CoV-2 Neutralizing Antibodies in blood samples
T-Cell Profile | Up to 24 months
  T-Cell Profile of blood samples

OTHER OUTCOMES:
Difference in Rates of Symptomatic COVID-19 Infection | Up to 24 Months
  Difference in rates of symptomatic COVID-19 infection following vaccination with mRNA SARS-CoV-2 vaccines between individuals with MS on B-cell depleting therapy and individuals with MS on non-cell depleting therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Strauss Farber, MD, Principal Investigator — Columbia University; Sarah Wesley, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No